CLINICAL TRIAL: NCT07022678
Title: A Randomized Double-Blinded Trial of Xylitol Dental Wipes for the Prophylaxis of Bloodstream Infections From Oral Organisms in Pediatric Patients With Acute Myeloid Leukemia
Brief Title: Xylitol Dental Wipes for the Reduction of Bloodstream Infection Risk in Children With Acute Myeloid Leukemia
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: ACCL2531; NCI-2025-03832 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ACCL2531 (Other: Children's Oncology Group); COG-ACCL2531 (Other: DCP); ACCL2531 (Other: CTEP); U24CA196173 (NIH); UG1CA189955 (NIH)
Record Dates: First submitted 2025-05-29; First posted 2025-06-15 (Actual); Last update posted 2025-08-18 (Actual); Status verified 2025-08

CONDITIONS: Acute Myeloid Leukemia; Recurrent Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Practice Guidelines as Topic; Standard of Care; Specimen Handling; Cytarabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The subject, investigators, and site-specific research and clinical staff who are involved with the conduct of the study will remain blinded to the treatment. The presence of a BSI event (either single organism or polymicrobial) will be determined by review of microbiology reports submitted to a central review committee whose members will be blinded to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm I (xylitol dental wipe) (Experimental): Patients receive standard chemotherapy containing cytarabine IV on study and receive a xylitol dental wipe intraorally BID to the teeth and gums at the start of the chemotherapy cycle and continuing for up to 30 days or until ANC >= 100/u/L following nadir. Treatment continues for 2 consecutive cycles of chemotherapy. Additionally, patients may optionally undergo saliva sample collections throughout the study.
  Interventions: Other: Best Practice; Procedure: Biospecimen Collection; Drug: Cytarabine; Other: Electronic Health Record Review; Other: Xylitol-containing Oral Wipe
- Arm II (non-xylitol dental wipe) (Active Comparator): Patients receive standard chemotherapy containing cytarabine IV on study and receive a non-xylitol dental wipe intraorally BID to the teeth and gums at the start of the chemotherapy cycle and continuing for up to 30 days or until ANC >= 100/u/L following nadir. Treatment continues for 2 consecutive cycles of chemotherapy. Additionally, patients may optionally undergo saliva sample collections throughout the study.
  Interventions: Other: Best Practice; Procedure: Biospecimen Collection; Drug: Cytarabine; Other: Electronic Health Record Review; Drug: Placebo Administration

INTERVENTIONS:
Other: Best Practice — Given standard chemotherapy
  Other Names: standard of care; standard therapy
Procedure: Biospecimen Collection — Undergo saliva sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Other: Electronic Health Record Review — Ancillary studies
Drug: Placebo Administration — Given intraorally
  Arms: Arm II (non-xylitol dental wipe)
Other: Xylitol-containing Oral Wipe — Given intraorally
  Other Names: Spiffies (TM) Xylitol Wipes; Xylitol Wipes
  Arms: Arm I (xylitol dental wipe)

SUMMARY:
This phase III trial compares the effect xylitol dental wipes to dental wipes without xylitol for the reduction of bloodstream infection in children with acute myeloid leukemia (AML). Xylitol is a naturally occurring sugar compound found in fruits and vegetables. Xylitol has been shown to limit the growth of bacteria in the mouth, and to reduce cavities, plaque on the teeth, and inflammation of the gums. Treatment for AML includes chemotherapy. Patients receiving chemotherapy for AML have a risk of developing bloodstream infections. Bloodstream infections can make patients very sick, can contribute to delays in treatment, and can even cause death. In AML patients, bacteria or fungus (yeast) can sometimes enter the bloodstream from the mouth. Using xylitol dental wipes may help to reduce bloodstream infections in children being treated for AML.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the incidence rate of bloodstream infections (BSI) (BSI per 1000 patient-days) from oral organisms over 2 cycles of chemotherapy in children with acute myeloid leukemia (AML) randomized to xylitol-containing oral wipes (xylitol dental wipes) versus control wipes.

SECONDARY OBJECTIVE:

I. To compare the rate of BSI (BSI per 1000 patient-days) from any organism in patients randomized to xylitol dental wipes versus control wipes.

EXPLORATORY OBJECTIVES:

I. To compare the frequency of severe infection (defined as any infection or infestation falling under Common Terminology Criteria for Adverse Events [CTCAE] sepsis grade 4 or 5) in patients randomized to xylitol dental wipes versus control wipes.

II. To compare the frequency of fever and neutropenia episodes in patients randomized to xylitol dental wipes versus control wipes.

III. To compare the frequency of severe mucositis, using the Children's International Mucositis Evaluation Scale (ChIMES), in patients randomized to xylitol dental wipes versus control wipes in addition to CTCAE grade 3 and above mucositis.

IV. To evaluate changes in oral microbial composition in pediatric patients treated with xylitol versus control wipes.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive standard chemotherapy containing cytarabine intravenously (IV) on study and receive a xylitol dental wipe intraorally twice daily (BID) to the teeth and gums at the start of the chemotherapy cycle and continuing for up to 30 days or until absolute neutrophil count (ANC) >= 100/u/L following nadir. Treatment continues for 2 consecutive cycles of chemotherapy. Additionally, patients may optionally undergo saliva sample collections throughout the study.

ARM II: Patients receive standard chemotherapy containing cytarabine IV on study and receive a non-xylitol dental wipe intraorally BID to the teeth and gums at the start of the chemotherapy cycle and continuing for up to 30 days or until ANC >= 100/u/L following nadir. Treatment continues for 2 consecutive cycles of chemotherapy. Additionally, patients may optionally undergo saliva sample collections throughout the study.

After completion of study treatment, patients are followed over the next cycle of chemotherapy or if chemotherapy is complete, for 90 days after the start of the last cycle of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be ≥ 1 year to ≤ 25 years old at enrollment.
* Patient must have a diagnosis of AML according to the 2016 World Health Organization classification with or without extramedullary disease. Patients with either newly diagnosed or relapsed AML are eligible as long as they meet the planned treatment criteria.
* Patient should be planned to receive at least 2 consecutive cycles of myelosuppressive chemotherapy. Each cycle must:

  * Contain IV cytarabine (liposomal formulations allowed), and
  * The duration of severe neutropenia should be expected to be ≥ 7 days. Hematopoietic stem cell transplantation (HSCT) conditioning cannot count as one of the two required planned cycles.

Note: Patients do not need to be co-enrolled on an upfront AML treatment protocol study, but co-enrollment is permitted.

* Minimum of one visible or erupted tooth.
* Agree to avoid xylitol containing gum or toothpaste during intervention period.
* All patients and/or their parents or legal guardians must sign a written informed consent.
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met.

Exclusion Criteria:

* Patients with Down syndrome-associated AML.
* Prior therapy: Prior radiation treatment for cancer of oral cavity, head or neck in past 6 months per study participant's medical record.
* Patients with known history of allergy to xylitol.
* Patients with known history of allergy to grapes or grape flavoring.
* Patients who are actively being treated for an oral organism related blood stream infection.
* Patients for whom the practitioner believes are unable to comply with use of oral dental wipes.

Ages: 1 Year to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 556 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2031-06-30 (Estimated); Study Completion 2032-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of bloodstream infections (BSI) from oral flora | Up to 37 days after the start date of the second cycle of chemotherapy that occurs while the patient is enrolled on study
  Will report the estimated oral organism BSI incidence rates by arm as number of events per 1000 patient-days. We will also report the incidence rate ratio under a Poisson regression model contrasting incidence rates of oral organism BSI for the treatment relative to control arm and the corresponding 95% confidence interval.

SECONDARY OUTCOMES:
Number of BSI from any organism | Up to 37 days after the start date of the second cycle of chemotherapy that occurs while the patient is enrolled on study
  Will report the estimated BSI incidence rates by arm as number of events per 1000 patient-days. We will also report the incidence rate ratio under a Poisson regression model contrasting incidence rates of BSI for the treatment relative to control arm and the corresponding 95% confidence interval.

OTHER OUTCOMES:
Severe infection (Common Terminology Criteria for Adverse Events (CTCAE) grade 4 or higher sepsis) | Up to 90 days after the start date of the second cycle of chemotherapy that occurs while the patient is enrolled on study
  Will report the proportion of patients who experience one or more episodes of febrile neutropenia while on study by arm as well as corresponding 95% confidence intervals.
Neutropenic fever episodes | Up to 90 days after the start date of the second cycle of chemotherapy that occurs while the patient is enrolled on study
  Will report the proportion of patients who experience one or more episodes of febrile neutropenia while on study by arm as well as corresponding 95% confidence intervals.
Severe mucositis (Common Terminology Criteria for Adverse Events (CTCAE) grade 3 or higher) | Up to 90 days after the start date of the second cycle of chemotherapy that occurs while the patient is enrolled on study
  Will report the proportion of patients who experience one or more episode of severe mucositis while on study by arm as well as corresponding 95% confidence intervals.
Oral microbial layout (as measured by beta diversity using the Bray-Curtis dissimilarity index) | Up to 42 days after the start date of the second cycle of chemotherapy that occurs while the patient is enrolled on study
  Will report the mean of Bray-Curtis dissimilarity index values by arm, using the final specimen (saliva) collection timepoint for each patient. Will report corresponding 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer J Wilkes, Principal Investigator — Children's Oncology Group